CLINICAL TRIAL: NCT01883804
Title: Open Label Pilot Study of the Effect of Methyldopa on MHC-II Antigen Presentation in Type 1 Diabetes
Brief Title: Effect of Methyldopa on MHC Class II Antigen Presentation in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1408
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Diabetes Mellitus; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Methyldopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): All participants selected to continue with Methyldopa administration.
  Interventions: Drug: Methyldopa

INTERVENTIONS:
Drug: Methyldopa — 6 weeks of Methyldopa administration; where the dose will be increased according to safety of efficacy.
  Other Names: Aldomet

SUMMARY:
Type 1 Diabetes is an autoimmune condition in which segments of the immune system cause the destruction of insulin producing cells in the pancreas, leaving individuals with an impaired ability to control blood glucose levels. Currently there is no cure for Type 1 Diabetes and the treatments involve lifelong insulin administration and careful monitoring of blood glucose levels. Long-term complications like cardiovascular disease, nerve damage, and retina damage, may result. Previous studies have shown that improvement in the control of blood glucose can reduce the risks from these long-term complications. Residual insulin production, typically within the first few years following diagnosis, helps to reduce an individual's need to supplement insulin by injection or pump. This effect helps in maintaining the body's ability to regulate blood glucose levels and reducing the needs of external insulin.

Methyldopa, or Aldomet, has been approved by the Food and Drug Administration and is commonly used to treat high blood pressure. This drug has been approved for several decades and has been shown to be safe and effective. This drug has been identified by the researcher to be able to block the communication between two important types of immune cells; which play a critical role in the autoimmune processes of Type 1 Diabetes. The investigators hypothesize that Methyldopa, over a 6 week treatment period, will block this communication and possibly slow down the destruction of insulin producing cells. The investigators hope to assess the appropriate and safe dose to achieve this effect, along with the drug's ability to maintain insulin production and blood glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes Mellitus
* 18-46 years of age
* Residual C-peptide production during screening
* Positive for at least one islet autoantibody: insulin (if only insulin autoantibody positive, determination must be within two weeks of insulin initiation), GAD-65, IA-2 or ZnT8
* Positive for at least one gene encoding HLA-DQ8 (DQB*0302)
* No history of difficult to control hypertension (defined as requiring > 2 anti-hypertensive medications)
* Agree to intensive management of diabetes with an HgbA1c goal of < 8.0%
* If female: (a) surgically sterile or (b) postmenopausal or (c) if of reproductive potential, willing to use medically acceptable birth control (e.g. female hormonal contraception, barrier methods or sterilization.) until study completion
* If male and of reproductive potential, willing to use medically acceptable birth control until study completion, unless the female partner is postmenopausal or surgically sterile

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the study protocol
* No HLA-DQ8 gene (DQB*0302)
* Difficult to control hypertension (defined as requiring > 2 anti-hypertensive medications)
* History of postural hypotension or Addison's disease
* Body Mass Index (BMI) > 30 kg/m2
* Unstable blood sugar control defined as one or more episodes of severe hypoglycemia (defined as hypoglycemia that required the assistance of another person) within the last 30 days
* Administration of an experimental agent for T1D at any time or use of an experimental device for T1D within 30 days of screening, unless approved by the study PI
* History of any organ transplant, including islet cell transplant
* Active autoimmune or immune deficiency disorder (e.g. sarcoidosis, rheumatoid arthritis)
* Anticipated pregnancy during the 12 week study period
* Any social or medical condition that would, in the opinion of the investigator, prevent complete participation in the study or that would pose a significant hazard to the subjects' participation
* History of active substance abuse within 12 months of screening
* A psychiatric or medical disorder that would prevent giving informed consent

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Michels, MD, Principal Investigator — Barbara Davis Center for Diabetes, University of Colorado School of Medicine
Locations (1):
- Barbara Davis Center for Diabetes, University of Colorado School of Medicine, Aurora, Colorado, United States

REFERENCES:
- [Result] Ostrov DA, Alkanani A, McDaniel KA, Case S, Baschal EE, Pyle L, Ellis S, Pollinger B, Seidl KJ, Shah VN, Garg SK, Atkinson MA, Gottlieb PA, Michels AW. Methyldopa blocks MHC class II binding to disease-specific antigens in autoimmune diabetes. J Clin Invest. 2018 May 1;128(5):1888-1902. doi: 10.1172/JCI97739. Epub 2018 Apr 3. PMID 29438107
- [Derived] Ostrov DA, Gottlieb PA, Michels AW. Rationally designed small molecules to prevent type 1 diabetes. Curr Opin Endocrinol Diabetes Obes. 2019 Apr;26(2):90-95. doi: 10.1097/MED.0000000000000470. PMID 30694829
- See also: Barbara Davis Center Website — http://www.barbaradaviscenter.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the adult clinic of the Barbara Davis Center, University of Colorado School of Medicine. Recruitment began in July of 2013 and concluded in November of 2015.
Pre-assignment Details: A total of 30 participants joined the study. Five participants withdrew prior to the first visit or any study procedures. The remaining 25 participants started the study and 20 completed all study visits and procedures.
Groups:
- Methyldopa Group: All participants selected to continue with Methyldopa administration.
  Methyldopa: 6 weeks of Methyldopa administration; where the dose will be increased according to safety of efficacy.
Period: Overall Study
Arm/Group | Methyldopa Group
Started | 25
Completed | 20
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Analysis population includes those participants that completed the course of the study.
Arm/Group | Study Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years]
  Mean Age | 24.75 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Duration of Type 1 Diabetes [Mean (Full Range); unit: Days] | 133 [21 to 566]
Hemoglobin A1c [Mean (Full Range); unit: Percentage] | 7.4 [5.3 to 12.1]
C-Peptide AUC following a 2 Hour Mixed Meal Tolerance Test [Mean (Full Range); unit: nmol/L/Min] | 0.64 [0.10 to 2.67]
Positive Insulin Autoantibodies (Index) [Count of Participants; unit: Participants] — Only included if measured within 21 days of starting exogenous insulin.
  Participants | 1
Positive GAD Autoantibodies [Count of Participants; unit: Participants] | 15
Positive IA-2 Autoantibodies [Count of Participants; unit: Participants] | 14
Positive ZnT8 Autoantibodies [Count of Participants; unit: Participants] | 11
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 113.2 (10.03)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 69.65 (8.16)
Elevated AST Values [Count of Participants; unit: Participants] | 0
Elevated ALT Values [Count of Participants; unit: Participants] | 0
Abnormal Hemoglobin Levels [Count of Participants; unit: Participants] — Hemoglobin < 12 g/dL
  Participants | 0

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline of DQ8 Antigen Presentation by Peripheral Blood Mononuclear Cells After 6 Weeks of Methyldopa Treatment.
Description: Cryopreserved primary peripheral blood mononuclear cells were used as antigen presenting cells to stimulate engineered T-cells (T-cell receptor transductant) responding to a specific peptide presented by HLA-DQ8. Secreted IL-2 from the engineered T-cell was measured by a highly sensitive ELISA. This was done for both an α-gliadin/DQ8 responding T-cell and a separate insulin/DQ8 responding T-cell.
Time Frame: 6 Weeks (Baseline and week 6)
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Groups:
- Study Group: open label treatment; dose escalation of methyldopa
Arm/Group | Study Group
Number analyzed (Participants) | 20
pg/mL
  Baseline, α-gliadin/DQ8 | 642 (104)
  6 weeks of treatment, α-gliadin/DQ8 | 430 (70)
  Baseline, insulin/DQ8 | 27.4 (5.2)
  6 weeks of treatment, insulin/DQ8 | 17.9 (3.3)

2. Secondary Outcome: The Change in C-Peptide AUC Following a MMTT From Baseline to Study Completion.
Description: Investigators aim to observe changes in residual endogenous insulin production as measured by C-peptide 2 hour area under the curve following a Mixed Meal Tolerance Test (MMTT). C-peptide is a measure of endogenous insulin secretion as both are secreted in a 1:1 molar ratio. Individuals ingested a liquid meal (Boost) with a fixed amount of protein, fat and carbohydrate in the fasting state followed by the timed measurements of serum C-peptide at 0, 15, 30, 60, 90 and 120 minutes to compute the AUC.
Time Frame: 12 weeks (Baseline and week 12)
Measure: Mean (Standard Deviation); unit: nmol/L/min
Arm/Group | Study Group
Number analyzed (Participants) | 20
nmol/L/min
  Baseline | 0.6 (0.5)
  Study Completion | 0.7 (0.6)

3. Secondary Outcome: The Change in Hemoglobin A1c From Baseline to Study Completion.
Description: Investigators aim to observe changes in hemoglobin A1c values, a measure of average blood glucose over the preceding 3 months.
Time Frame: 12 weeks (Baseline and week 12)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Study Group
Number analyzed (Participants) | 20
percentage
  Baseline | 7.4 (1.6)
  Study Completion | 6.5 (0.8)

4. Secondary Outcome: The Change in Insulin Use From Baseline to Study Completion.
Description: Exogenous insulin use per kg of body weight.
Time Frame: 12 weeks (Baseline and week 12)
Measure: Mean (Standard Deviation); unit: units/Kg body weight
Arm/Group | Study Group
Number analyzed (Participants) | 20
units/Kg body weight
  Baseline | 0.37 (0.20)
  Study Completion | 0.36 (0.19)

ADVERSE EVENTS:
Time Frame: Over the course of the 12 week study.
Description: Adverse event collection occurred at each visit through standard questions asked by the research coordinator and discussions with the investigator.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 5/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=25)
Fatigue (General disorders) | 5 (5) — A state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities. Grade 2 are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No